CLINICAL TRIAL: NCT03832660
Title: Clinical and Genetic Determinants of Disease Progression and Response to Sacubitril/Valsartan vs Lifestyle (Physical Activity and Dietary Nitrate) in Patients With Hypertrophic Cardiomyopathy
Brief Title: Sacubitril/Valsartan vs Lifestyle in Hypertrophic Cardiomyopathy
Acronym: SILICOFCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); University Hospital Regensburg (Other); Institute of Cardiovascular Diseases, Vojvodina (Other); University of Belgrade (Other)
Responsible Party: Principal Investigator, Djordje Jakovljevic, Senior Lecturer/Associate Professor in Cardiovascular Ageing and Heart Failure, Newcastle University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252015
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Lifestyle; ARNI; Exercise tolerance
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lifestyle (Active Comparator): Lifestyle intervention will consist of two integrated components i.e. physical activity and dietary supplementation with inorganic nitrate. The physical activity component aims to increase daily physical activity level by at least 2000 steps/day from baseline (e.g. walking for approximately 30 minutes), at least 5-7 days per week. The second component of the lifestyle intervention is a dietary supplementation with inorganic nitrate. A single dose of inorganic nitrate given in the form of concentrated nitrate-rich beetroot juice (NO3-, BEET IT Sport, James White Drinks Ltd., Ipswich, UK) containing 6 mmol of NO3- in 70 ml bottle.
  Interventions: Behavioral: Lifestyle
- Sacubitril/Valsartan (Active Comparator): Sacubitril / Valsartan as a pharmacological agent shall be studied to verify its effects on cardiac morphology and physiology of hypertrophic cardiomyopathy patients.
  Interventions: Drug: Sacubitril/Valsartan
- Usual Care (No Intervention): The participants in control group do not undertake lifestyle or sacubitril / valsartan intervention.

INTERVENTIONS:
Behavioral: Lifestyle — A 4-month lifestyle intervention will consist of two integrated components i.e. physical activity and dietary supplementation with inorganic nitrate. The physical activity component aims to increase daily physical activity level by at least 2000 steps/day from baseline (e.g. walking for approximately 30 minutes), at least 5-7 days per week. The second component of the lifestyle intervention is a dietary supplementation with inorganic nitrate. A single dose of inorganic nitrate given in the form of concentrated nitrate-rich beetroot juice (NO3-, BEET IT Sport, James White Drinks Ltd., Ipswich, UK) containing 6 mmol of NO3- in 70 ml bottle.
  Other Names: Physical acitivity and dietary nitrate
  Arms: Lifestyle
Drug: Sacubitril/Valsartan — Angiotensin receptor neprilysin inhibitor Sacubitril / Valsartan: The treatment period begins on day 1 with initial dosing of sacubitril/valsartan, followed by uptitration every 2 to 4 weeks to the target dose of 97/103 mg twice daily. 3 doses of sacubitril/valsartan available throughout the study are 24/26 mg, 49/51 mg, and 97/103 mg, each taken by mouth twice daily. If the patient discontinues the study medication, the patient is advised to return to the clinic for an end-of-study visit. Patients undergo treatment for 4 months.
  Other Names: Pharmacological
  Arms: Sacubitril/Valsartan

SUMMARY:
The overall aim of this project is to establish potential benefits of a novel lifestyle (physical activity and dietary nitrate) and pharmacological (angiotensin receptor neprilysin inhibitor) interventions in patients with hypertrophic cardiomyopathy (HCM). HCM is the most common genetic cardiovascular disease with a broad spectrum of disease severity. Angiotensin receptor neprilysin inhibitor reduces death, hospitalisation, and may improve cardiac function and exercise tolerance in heart failure. Exercise training is associated with a significant increase in exercise tolerance, but appear to have limited effect on measures of cardiac morphology or function in patients with HCM. Dietary supplementation with inorganic nitrate (i.e. concentrated nitrate-rich beetroot juice) improves exercise capacity, vasodilatation and cardiac output reserves while reduces arterial wave reflections, which are linked to left ventricular diastolic dysfunction and remodelling. Using a five-centre, open label, three-arm, pilot design, the present study will evaluate the effect of lifestyle (physical activity and dietary supplementation with inorganic nitrate) and pharmacological (angiotensin receptor neprilysin inhibitor sacubitril / valsartan) interventions in patients with HCM. The Aim is to examine whether these interventions improve functional capacity, clinical phenotypic characteristics, and quality of life in patients with HCM.

DETAILED DESCRIPTION:
Background and Rationale for the Study:

Hypertrophic cardiomyopathy (HCM) is the most common hereditary cardiac disease, affecting one in 500 individuals. The predominant cause is mutation of genes that encode protein components of the cardiac sarcomere. The mechanisms that lead from a sarcomere gene mutation to phenotypic expression of HCM are poorly understood, which impedes the search for a treatment that can disrupt the pathophysiological process.

The clinical diagnosis of HCM is based on hypertrophy of the left ventricle that cannot be explained by extrinsic factors such as increased afterload. The course of the disease is highly variable, ranging from an asymptomatic, benign course with a normal life expectancy to a progressive disease characterised by angina, heart failure, atrial fibrillation, stroke, malignant arrhythmia, syncope, or sudden cardiac death. Disease progression can relate to increasing left ventricular hypertrophy and fibrosis leading to worsening of diastolic (and occasionally systolic) function, increased left ventricular end-diastolic pressure, and left atrial enlargement. No medical treatment has been reliably shown to halt or reverse disease progression. Clinical trials demonstrated limited or no effect of angiotensin receptor blockers or late sodium current inhibitor on disease progression, cardiac structure and function, exercise tolerance and quality of life in patients with HCM. Accordingly, treatment recommendations are focused on the alleviation of symptoms, prevention of thromboembolic events, and implantation of prophylactic implantable cardioverter defibrillators in patients at high risk of sudden cardiac death.

Lifestyle interventions including physical activity and dietary nitrate supplementation are safe and can improve symptoms and signs in patients with heart failure. Exercise training is associated with a significant increase in exercise tolerance, but appear to have limited effect on measures of cardiac morphology or function in patients with HCM. Dietary supplementation with inorganic nitrate (i.e. concentrated nitrate-rich beetroot juice) improves exercise capacity, vasodilatation and cardiac output reserves while reduces arterial wave reflections, which are linked to a left ventricular diastolic dysfunction and remodelling.

Angiotensin receptor neprilysin inhibitor (ARNI) is a novel treatment shown to reduce mortality and hospitalisation in heart failure with reduced ejection fraction, while there is an ongoing trial to evaluate its effect on heart failure with preserved ejection fraction. Recent preliminary data suggest that ARNI improves left ventricular wall motion and exercise tolerance, while reduces markers of left ventricular wall stress. The impact of ARNI on parameters of cardiac function and remodeling has not been previously described in heart failure. Several trials are ongoing aiming provide mechanistic insight on the effect of ARNI in heart failure. The effect of ARNI has not been evaluated in patients with HCM.

Despite both lifestyle and ARNI interventions may have potential positive effect, no study so far has evaluated their effect on exercise tolerance, cardiac remodelling and quality of life in patients with HCM.

Aim and Objectives:

The aim of the project is to identify clinical and genetic markers of disease progression and response to lifestyle and pharmacological interventions in patients with hypertrophic cardiomyopathy. Specifically, the project will examine whether i) Lifestyle intervention incorporating physical activity and dietary supplementation with inorganic nitrate, and ii) Angiotensin receptor neprilysin inhibitor, improve functional capacity, clinical phenotypic characteristics, and quality of life in patients with HCM.

Study Design and Methods:

The Investigators propose to study at least 240 patients across five centres using an open label, three-arm trial designed to evaluate the effect of lifestyle (physical activity and dietary supplementation with inorganic nitrate) and pharmacological intervention (angiotensin receptor neprilysin inhibitor sacubitril / valsartan) in patients with HCM who are currently not participating in any drug trial or a regular exercise regimen (i.e. ≤ minutes of exercise, ≤ 1 day per week for the previous 3 months). All patients will be administered a pre-screening questionnaire in order to determine eligibility and will be randomized into a intervention or a standard (control) care group in the 2:1 ratio. This will be a collaborative effort with investigators from Germany - University Hospital Regensburg (Dr Lars Maier), Italy - Azienda Ospedaliero Universitaria Careggi Florence (Dr Iacopo Olivotto), Serbia - Institute of Cardiovascular Diseases of Vojvodina (Dr Lazar Velicki), Serbia - University of Belgrade Faculty of Medicine (Drs Arsen Ristic and Dejana Popovic) and United Kingdom - University of Newcastle (Drs Djordje Jakovljevic and Guy MacGowan). Investigator will secure their own Ethics Committee / Institutional Review Board approvals. Target number is at least 45 patients at each centre.

Recruitment procedures:

Potentially eligible patients will be identified through the Cardiology clinics of the participating centres. Patients will be identified and contacted by the member of the study research team. An information sheet will be mailed out upon request. Consent forms will be signed by the participant and countersigned by a member of the study team during the first research visit.

Interventions:

Duration of the lifestyle and pharmacological interventions is four months.

Lifestyle Intervention:

The lifestyle intervention will consist of two integrated components i.e. physical activity and dietary supplementation with inorganic nitrate.

The first component of the lifestyle intervention is physical activity component is a validated home-based exercise intervention aiming to increase daily physical activity level by at least 2000 steps/day from baseline (e.g. walking for approximately 30 minutes), at least 5-7 days per week, as this increment in daily physical activity was associated with a 10% lower risk of a cardiovascular events in high risk patients.

To control for exercise intensity patients will be instructed to use standardised Borg Scale (0-20) to rate perceived exertion aiming for achieving the levels between 11 - 13 (easy-light-to somewhat hard). The exercise prescription will be progressed individually as conditioning takes place, with the emphasis placed on volume of activity i.e. duration before intensity. Targets will be set by participants, but the Investigators will present potential health benefits of increasing physical activity by 2000 steps per day at least five days per week (≥150 minutes per week). No strength training or burst activity will be prescribed and all activities will fall well within the recommended national guidelines for recreational exercise. Patients will be counselled to hydrate adequately during exercise, and to be alert to warning signs and symptoms that should prompt them to stop exercising and contact the research team. All patients will be provided with pedometers and asked to complete a daily physical activity diary which will be reviewed and discussed on a weekly basis (telephone call) with the member of the research team. All study patients will keep an exercise log and be provided with pedometers.

The second component of the lifestyle intervention is a dietary supplementation with inorganic nitrate. A single dose of inorganic nitrate given in the form of concentrated nitrate-rich beetroot juice (NO3-, BEET IT Sport, James White Drinks Ltd., Ipswich, UK) containing 6 mmol of NO3- in 70 ml bottle. Instructions will be provided for self-administration of the nutritional intervention and patients will be asked to consume beetroot juice each morning with the breakfast for 4 months.

The EPIC Food Frequency Questionnaire (FFQ) will be administered at baseline and the FETA software used to extract dietary (energy and nutrient) information. Adherence to the intervention will be tracked by completion of activity logs, weekly telephone follow-ups, pedometers, and self-reported diaries.

Pharmacological Intervention (Angiotensin receptor neprilysin inhibitor sacubitril / valsartan):

Patients who meet the study inclusion/exclusion criteria, after signing the informed consent, will be invited to the screening visit. Patients previously receiving angiotensin-converting enzyme inhibitor or angiotensin receptor blocker therapy will require a 36-hour washout period before initiation of sacubitril/valsartan to reduce the risk of angioedema.

The treatment period begins on day 1 with initial dosing of sacubitril/valsartan, followed by uptitration every 2 to 4 weeks, according to the prescribing information, to the target dose of 97/103 mg twice daily. The 3 doses of sacubitril/valsartan available throughout the study are 24/26 mg (dose level 1), 49/51 mg (dose Level 2), and 97/103 mg (dose Level 3), each taken by mouth twice daily.

Doses may be adjusted based on overall safety and tolerability. If necessary, dose adjustments or elimination of concomitant medications is made to alleviate adverse effects. If adverse effects are not alleviated or it is not possible to adjust concomitant medications, the study treatment may be down-titrated by 1 dose level-or, at the lowest dose, temporarily withdrawn-for 1 to 4 weeks. The patient may then be reassessed and the study treatment further down-titrated every 1 to 4 weeks until the patient is deemed stable. Once stability is achieved, the patient is re-challenged with up-titration to the target dose. If the patient discontinues the study medication, the patient is advised to return to the clinic for an end-of-study visit. Patients undergo treatment for four months.

Control group / Usual Care Patients with HCM typically do not receive exercise and/or nutritional therapies. The choice of a usual care (no intervention) comparator in this pilot study is therefore reflective of the situation for the vast majority of patients with HCM. In this study, the intervention and control group will receive usual medical management for HCM according to national and local guidelines. Patients in the control group will also be provided with activity logs, weekly telephone follow-ups, pedometers, and self-reported diaries but will be asked not to change their physical activity and dietary habits during the study.

Research Visits Eligible patients will attend the Clinical Research Facilities of five participating centres for the total of 5 visits i.e. two at baseline (Visit 1 and Visit 2), and two at 4-month (Visit 3 and Visit 4) when the assessments performed during Visits 1 and 3 (detailed below) will be repeated.

Patients will be given new activity logs at the end of 4-month protocol period and these logs will be reviewed 3 months later (7 months after study initiation) during the follow-up visit (Visit 5) During this visit patients will be asked to complete quality of life questionnaires. Additionally, physical activity will be reviewed and patients will be asked to repeat cardiopulmonary exercise test.

Patients will be contacted via email, telephone or spoken to in person to discuss the project and will be taken through the information sheet to ensure they understand the nature of the study.

The following testing will be performed at study initiation and termination:

1. Bloods, body composition, electrocardiography, cardiac autonomic function, arterial stiffness.
2. Cardiopulmonary exercise testing in combination with echocardiography.
3. Cardiac magnetic resonance imaging in patients without implantable devices.
4. Quality of life, Anxiety and Depression, and Food Frequency questionnaires.

Funding: This project has received funding from the European Union's Horizon 2020 Research and Innovation Programme under Grant Agreement no. 777204.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of obstructive and/or non-obstructive hypertrophic cardiomyopathy.
* Agreement to be a participant in the study protocol and willing/able to return for follow-up.
* Able to provide written informed consent

Exclusion Criteria:

* Less than 3 months post septal reduction therapy (surgery or catheter based intervention)
* Clinical decompensation in the previous 3 months, defined as New York Heart Association class IV congestive heart failure symptoms.
* Resting blood pressure greater than 180/100 mm Hg.
* Systolic blood pressure lower than 100 mmHg
* Hypotensive response to exercise testing (≥20 mmHg decrease of systolic blood pressure from baseline blood pressure or an initial increase in systolic blood pressure followed by a decrease of systolic blood pressure ≥20 mmHg).
* Use of angiotensin converting Enzyme inhibitors or angiotensin receptor blockers.
* Resting left ventricular outflow tract gradient > 50 mm Hg.
* Left ventricular ejection fraction of less than 50% by echocardiography.
* Implanted pacemaker or cardiodefibrilator in the last 3 months or scheduled.
* Renal insufficiency with a glomerular filtration rate of less than 30 mL/min per 1.73m2.
* Present or planned pregnancy.
* Life expectancy less than 12 months.
* Body mass index >40 kg/m2.
* A history of exercise induced syncope or ventricular arrhythmias.
* Inability to exercise due to orthopaedic or other non-cardiovascular limitations.
* Use of other investigational drugs at the time of enrolment.
* Any surgical or medical condition that in the opinion of the investigator may place the patient at higher risk from his/her participation in the study or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* History or presence of any other disease with a life expectancy of <3 years
* History of noncompliance to medical regimens and patients who are considered potentially unreliable.
* History or evidence of drug or alcohol abuse within the past 12 months.
* History of malignancy of any organ system (other than localized basal or squamous cell carcinoma of the skin or localized prostate cancer), treated or untreated, within the past 2 years, regardless of whether there is evidence of local recurrence or metastases.
* Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and AF or atrial flutter with a resting ventricular rate >110 beats per minute.
* Participation in competitive or organized sport activities (such as football, basketball, rugby, hockey, etc), burst activity (such as sprinting, racket sports, etc) or heavy isometric exercise (such as body building or bench-pressing) or opposition of refraining from the same for the duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (ml/kg/min) | 4 months
  Change in exercise tolerance i.e. peak oxygen consumption and anaerobic threshold post intervention

SECONDARY OUTCOMES:
Left ventricular mass (grams) | 4 months
  The size of the left ventricle
LVOT obstruction | 4 months
  Degree of left ventricular outflow tract obstruction.
LVEF (%) | 4 months
  Left ventricular ejection fraction
Minnesota Living with Heart Failure questionnaire | 4 months
  Quality of Life (score range from 0 to 105)
SF36 questionnaire | 4 months
  Quality of Life RAND 36-Item Health Survey (score range from 0 to 100)
E/A ratio | 4 months
  Early to late filling ratio

CONTACTS AND LOCATIONS:
Overall Officials: Dr Djordje G Jakovljevic, Principal Investigator — Newcastle University Faculty of Medical Sciences, Clinical Research Facility, Newcastle upun Tyne Hospitals NHS Foundation Trust
Locations (5):
- University Hospital Regensburg, Regensburg, Germany
- Azienda Ospedaliero Universitaria Careggi Florence, Florence, Italy
- Serbia (2):
  - University of Belgrade Faculty of Medicine, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
- Newcastle University, Faculty of Medical Sciences, Clinical Research Facility, Royal Victoria Infirmary; Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual patient data will be shared between the partners of the SILICOFCM project.
Supporting Information: Study Protocol
Time Frame: January 2022, for five years
Access Criteria: Data will be available upon request to a principal investigator.
URL: http://silicofcm.eu

REFERENCES:
- [Result] Maron BJ, Gardin JM, Flack JM, Gidding SS, Kurosaki TT, Bild DE. Prevalence of hypertrophic cardiomyopathy in a general population of young adults. Echocardiographic analysis of 4111 subjects in the CARDIA Study. Coronary Artery Risk Development in (Young) Adults. Circulation. 1995 Aug 15;92(4):785-9. doi: 10.1161/01.cir.92.4.785. PMID 7641357
- [Result] Morita H, Rehm HL, Menesses A, McDonough B, Roberts AE, Kucherlapati R, Towbin JA, Seidman JG, Seidman CE. Shared genetic causes of cardiac hypertrophy in children and adults. N Engl J Med. 2008 May 1;358(18):1899-908. doi: 10.1056/NEJMoa075463. Epub 2008 Apr 9. PMID 18403758
- [Result] Force T, Bonow RO, Houser SR, Solaro RJ, Hershberger RE, Adhikari B, Anderson ME, Boineau R, Byrne BJ, Cappola TP, Kalluri R, LeWinter MM, Maron MS, Molkentin JD, Ommen SR, Regnier M, Tang WH, Tian R, Konstam MA, Maron BJ, Seidman CE. Research priorities in hypertrophic cardiomyopathy: report of a Working Group of the National Heart, Lung, and Blood Institute. Circulation. 2010 Sep 14;122(11):1130-3. doi: 10.1161/CIRCULATIONAHA.110.950089. No abstract available. PMID 20837938
- [Result] Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2011 Dec 13;58(25):2703-38. doi: 10.1016/j.jacc.2011.10.825. Epub 2011 Nov 8. No abstract available. PMID 22075468
- [Result] Maron BJ, Casey SA, Hauser RG, Aeppli DM. Clinical course of hypertrophic cardiomyopathy with survival to advanced age. J Am Coll Cardiol. 2003 Sep 3;42(5):882-8. doi: 10.1016/s0735-1097(03)00855-6. PMID 12957437
- [Result] Shimada YJ, Passeri JJ, Baggish AL, O'Callaghan C, Lowry PA, Yannekis G, Abbara S, Ghoshhajra BB, Rothman RD, Ho CY, Januzzi JL, Seidman CE, Fifer MA. Effects of losartan on left ventricular hypertrophy and fibrosis in patients with nonobstructive hypertrophic cardiomyopathy. JACC Heart Fail. 2013 Dec;1(6):480-7. doi: 10.1016/j.jchf.2013.09.001. Epub 2013 Oct 24. PMID 24621999
- [Result] Axelsson A, Iversen K, Vejlstrup N, Ho C, Norsk J, Langhoff L, Ahtarovski K, Corell P, Havndrup O, Jensen M, Bundgaard H. Efficacy and safety of the angiotensin II receptor blocker losartan for hypertrophic cardiomyopathy: the INHERIT randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2015 Feb;3(2):123-31. doi: 10.1016/S2213-8587(14)70241-4. Epub 2014 Dec 19. PMID 25533774
- [Result] Olivotto I, Camici PG, Merlini PA, Rapezzi C, Patten M, Climent V, Sinagra G, Tomberli B, Marin F, Ehlermann P, Maier LS, Fornaro A, Jacobshagen C, Ganau A, Moretti L, Hernandez Madrid A, Coppini R, Reggiardo G, Poggesi C, Fattirolli F, Belardinelli L, Gensini G, Mugelli A. Efficacy of Ranolazine in Patients With Symptomatic Hypertrophic Cardiomyopathy: The RESTYLE-HCM Randomized, Double-Blind, Placebo-Controlled Study. Circ Heart Fail. 2018 Jan;11(1):e004124. doi: 10.1161/CIRCHEARTFAILURE.117.004124. PMID 29321131
- [Result] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Result] Solomon SD, Rizkala AR, Gong J, Wang W, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Shi VC, Lefkowitz MP, McMurray JJV. Angiotensin Receptor Neprilysin Inhibition in Heart Failure With Preserved Ejection Fraction: Rationale and Design of the PARAGON-HF Trial. JACC Heart Fail. 2017 Jul;5(7):471-482. doi: 10.1016/j.jchf.2017.04.013. Epub 2017 Jun 26. PMID 28662936
- [Result] Beltran P, Palau P, Dominguez E, Faraudo M, Nunez E, Guri O, Mollar A, Sanchis J, Bayes-Genis A, Nunez J. Sacubitril/valsartan and short-term changes in the 6-minute walk test: A pilot study. Int J Cardiol. 2018 Feb 1;252:136-139. doi: 10.1016/j.ijcard.2017.10.074. PMID 29249422
- [Result] Solomon SD, Zile M, Pieske B, Voors A, Shah A, Kraigher-Krainer E, Shi V, Bransford T, Takeuchi M, Gong J, Lefkowitz M, Packer M, McMurray JJ; Prospective comparison of ARNI with ARB on Management Of heart failUre with preserved ejectioN fracTion (PARAMOUNT) Investigators. The angiotensin receptor neprilysin inhibitor LCZ696 in heart failure with preserved ejection fraction: a phase 2 double-blind randomised controlled trial. Lancet. 2012 Oct 20;380(9851):1387-95. doi: 10.1016/S0140-6736(12)61227-6. Epub 2012 Aug 26. PMID 22932717
- [Result] Januzzi JL, Butler J, Fombu E, Maisel A, McCague K, Pina IL, Prescott MF, Riebman JB, Solomon S. Rationale and methods of the Prospective Study of Biomarkers, Symptom Improvement, and Ventricular Remodeling During Sacubitril/Valsartan Therapy for Heart Failure (PROVE-HF). Am Heart J. 2018 May;199:130-136. doi: 10.1016/j.ahj.2017.12.021. Epub 2018 Feb 13. PMID 29754651
- [Result] Saberi S, Wheeler M, Bragg-Gresham J, Hornsby W, Agarwal PP, Attili A, Concannon M, Dries AM, Shmargad Y, Salisbury H, Kumar S, Herrera JJ, Myers J, Helms AS, Ashley EA, Day SM. Effect of Moderate-Intensity Exercise Training on Peak Oxygen Consumption in Patients With Hypertrophic Cardiomyopathy: A Randomized Clinical Trial. JAMA. 2017 Apr 4;317(13):1349-1357. doi: 10.1001/jama.2017.2503. PMID 28306757
- [Result] Zamani P, Rawat D, Shiva-Kumar P, Geraci S, Bhuva R, Konda P, Doulias PT, Ischiropoulos H, Townsend RR, Margulies KB, Cappola TP, Poole DC, Chirinos JA. Effect of inorganic nitrate on exercise capacity in heart failure with preserved ejection fraction. Circulation. 2015 Jan 27;131(4):371-80; discussion 380. doi: 10.1161/CIRCULATIONAHA.114.012957. Epub 2014 Dec 22. PMID 25533966
- [Result] Chirinos JA, Londono-Hoyos F, Zamani P, Beraun M, Haines P, Vasim I, Varakantam S, Phan TS, Cappola TP, Margulies KB, Townsend RR, Segers P. Effects of organic and inorganic nitrate on aortic and carotid haemodynamics in heart failure with preserved ejection fraction. Eur J Heart Fail. 2017 Nov;19(11):1507-1515. doi: 10.1002/ejhf.885. Epub 2017 May 25. PMID 28547861
- [Result] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Result] Yates T, Haffner SM, Schulte PJ, Thomas L, Huffman KM, Bales CW, Califf RM, Holman RR, McMurray JJ, Bethel MA, Tuomilehto J, Davies MJ, Kraus WE. Association between change in daily ambulatory activity and cardiovascular events in people with impaired glucose tolerance (NAVIGATOR trial): a cohort analysis. Lancet. 2014 Mar 22;383(9922):1059-66. doi: 10.1016/S0140-6736(13)62061-9. Epub 2013 Dec 20. PMID 24361242
- [Result] Mulligan AA, Luben RN, Bhaniani A, Parry-Smith DJ, O'Connor L, Khawaja AP, Forouhi NG, Khaw KT; EPIC-Norfolk FFQ Study. A new tool for converting food frequency questionnaire data into nutrient and food group values: FETA research methods and availability. BMJ Open. 2014 Mar 27;4(3):e004503. doi: 10.1136/bmjopen-2013-004503. PMID 24674997

DOCUMENTS (1):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03832660/Prot_000.pdf